CLINICAL TRIAL: NCT01292512
Title: Bereavement Management. Description, Assessment and Care. A Randomized Controlled Study.
Brief Title: Bereavement Management - Description, Assessment and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Dæhnfeldt Foundation (Unknown); TrygFonden, Denmark (Industry); Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Bereavement Management.
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2012-03

CONDITIONS: Bereavement; Grief
Keywords: Bereavement management; Complicated grief

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): A) Professional level. B) Patient level.
  Intervention
  Professional level:
  General Practitioners (GP) receive updated information on bereavement related symptoms, how to identify complicated grief, and the Dual Process Model (DPM) of coping.
  GPs receive suggestions on how to provide psycho-educational support for the patient.
  GPs are informed about the results of the initial assessment of their patient prognostic screening for complicated grief.
  Patient level:
  Patients receive updated information on bereavement related symptoms, the DPM of coping and suggestions on when to seek professional help.
  Patients are informed of the results of their initial assessment of their prognostic grief screening.
  Patients are encouraged to contact their GP if they worry about handling their bereavement reaction.
  Interventions: Other: Prognostic screening for complicated grief
- Control group (Other): Treatment as usual (in the Danish health care system).
  Interventions: Other: Prognostic screening for complicated grief

INTERVENTIONS:
Other: Prognostic screening for complicated grief — Patients in the intervention group are prognostically screened for development of complicated grief to identify those in need of help.

SUMMARY:
This study aims to develop a risk assessment tool to identify bereaved in risk of complicated grief reactions and to implement a bereavement management programme in primary health care based on the Dual Process Model of coping with bereavement. Furthermore to enhance bereavement care in general practice and to enhance patients' self-management in bereavement care.

DETAILED DESCRIPTION:
In Denmark alone there are approximately 55.000 deaths annually which leave approximately 200.000 bereaved close relatives. International studies show that 10-15% of bereaved persons develop complications following the death of a close relative. If those studies hold true, approximately 20 - 30.000 individuals annually will develop complications as a result of suffering a loss, and there is hardly any knowledge of how bereavement is treated or even legitimized in primary care and referred on to specialized (psychological or psychiatric) care. The field of bereavement is in need of studies that validate the theoretical underpinnings of the research area, enhanced assessment of predictive risk factors and updated intervention methods: in short a scientifically valid management programme.

ELIGIBILITY:
Inclusion Criteria:

* Newly bereaved from one of the inclusion facilities.
* 18 years or older.
* Danish citizen.
* Able to understand and speak Danish.
* Informed consent.
* Mentally able to cooperate

Exclusion Criteria:

* Patients with known substance abuse.
* Patients with recently (within 5 years) diagnosed psychopathological disorders that trigger psychotic episodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effect of the intervention measured by an increase in the diagnosis of complicated grief. | 20 months
  GPs receive updated information on bereavement related symptoms, how to identify complicated grief, and the Dual Process Model of coping.

SECONDARY OUTCOMES:
Effect of the intervention measured by register-based data. | 20 months
  Effect of the intervention measured by register-based data on frequency in contact with GP, referrals to psychological/psychiatric counselling, medicine consumption and use of emergency services.

CONTACTS AND LOCATIONS:
Overall Officials: Frede Olesen, Professor, Study Chair — Research Unit for General Practice, Aarhus University, Denmark
Locations (1):
- Research Unit for General Practice, Aarhus, Denmark

REFERENCES:
- [Derived] Guldin MB, Vedsted P, Jensen AB, Olesen F, Zachariae R. Bereavement care in general practice: a cluster-randomized clinical trial. Fam Pract. 2013 Apr;30(2):134-41. doi: 10.1093/fampra/cms053. Epub 2012 Sep 10. PMID 22964078